CLINICAL TRIAL: NCT04483037
Title: Comparison of Same-Day and Split-Dose Preparation With Sodium Picosulfate/Magnesium Citrate (Bowklean) for Afternoon Colonoscopy: A Randomized Non-Inferiority Study
Brief Title: Different Dosing Time of Bowklean for the Bowel Preparation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Changhua Christian Hospital (Other)
Responsible Party: Principal Investigator, HSUHENG YEN, Head of Endoscopy Room, Changhua Christian Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: CCH IRB No.: 181216
Record Dates: First submitted 2020-07-20; First posted 2020-07-23 (Actual); Last update posted 2021-07-23 (Actual); Status verified 2021-07

CONDITIONS: Bowel Preparation

STUDY DESIGN:
Intervention Model Description: The 1st group: split dose, day before, colonoscopy in the morning. The 2nd group: split dose, day before, colonoscopy in the afternoon. The 3rd group: same day, colonoscopy in the afternoon.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- split dose, day before, colonoscopy in the morning (Observation Group) (Active Comparator): routine bowel preparation before colonoscopy in the morning
  Interventions: Drug: Bowklean
- split dose, day before, colonoscopy in the afternoon (Random) (Active Comparator): routine bowel preparation before colonoscopy in the afternoon
  Interventions: Drug: Bowklean
- two dose in the same day, colonoscopy in the afternoon (Random) (Experimental): experimental group
  Interventions: Drug: Bowklean

INTERVENTIONS:
Drug: Bowklean — assigned intervention

SUMMARY:
The primary objective of this study is to compare the efficacy of administration routine bowel cleansing medication (Bowklean) for the Bowel Preparation at Different Times Prior Colonoscopy in the morning or in the afternoon.

DETAILED DESCRIPTION:
Sodium picosulfate/magnesium citrate (SPMC) is a small-volume bowel cleansing agent with similar efficacy and better tolerability than polyethylene glycol. However, there was limited data about the bowel cleansing efficacy of SPMC in comparing the same-day and split-dose preparation for afternoon colonoscopy.

This randomized, single-center, endoscopist-blinded, non-inferior study compared same-day (101 subjects) and split-dose (96 subjects) preparation with SPMC for afternoon colonoscopy. One additional prospective observation group of 100 subjects receiving colonoscopy in the morning was included as an observation group to compare bowel preparation in morning and afternoon colonoscopy. Efficacy of bowel cleansing was evaluated by the Aronchick Scale, Ottawa Bowel Preparation Scale (OBPS), Boston Bowel Preparation Scale (BBPS), and the Bubble Scale (TBS).

ELIGIBILITY:
Inclusion Criteria:

1. Subject is 20 and 99 years, inclusive.
2. Men or non-pregnant women who are scheduled for an elective colonoscopy.
3. Subjects should be willing, able to complete the entire procedure and to comply with study instructions.
4. Written informed consent obtained prior to study.

Exclusion Criteria:

1. Patients who are not suitable for colonoscopy

   * Acute surgical abdominal conditions (e.g. acute obstruction or perforation, etc.)
   * Active (acute/exacerbation of/severe/uncontrolled) Inflammatory Bowel Disease (IBD)
   * Colon disease (history of colonic cancer, toxic megacolon, toxic colitis, idiopathic pseudo- obstruction, hypomotility syndrome)
   * Gastrointestinal disorder (active ulcer, outlet obstruction, gastric retention, gastroparesis, ileus)
   * Uncontrolled angina and/or Myocardial Infarction (MI) within last 3 months before randomization, Congestive Heart Failure (CHF), arrhythmia, cardiomyopathy or uncontrolled hypertension
   * Renal insufficiency
2. Any prior colorectal surgery

   * in the past 3 months, excluding appendectomy, hemorrhoid surgery or prior endoscopic procedures
   * History of upper gastrointestinal surgery (gastric resection, gastric banding, gastric by-pass)
3. Severe chronic constipation
4. Hypersensitivity to any ingredient in the study medication

Ages: 20 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 297 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Aronchick Scale Bowel Cleaning Scale | during colonoscopy
  Aroochick Scale ranges from score 1 : excellent, 2: good, 3: fair, 4: poor 5: failed

SECONDARY OUTCOMES:
Boston Bowel Preparation Scale (BBPS) Bowel Cleaning Scale | During Colonoscopy
  The Boston Bowel Preparation Scale Score 0 : inadequate ; Score 1: fair ;Score 2: good; Score 3: excellent . min : 0 , max: 3
Colonscopy Bubble Scale | During Colonoscopy
  Colon Bubble Scale : Grade A : no bubble , Grade B: little bubble , Grade C: bubble of half of the lumen , Grade D: bubble of entire lumen. Grade A means the best and Grade D means the worst.

CONTACTS AND LOCATIONS:
Overall Officials: HsuHeng Yen, MD, Principal Investigator — Changhua Christian Hospital
Locations (1):
- Hsu-Heng Yen, Changhua, Taiwan

IPD SHARING:
Plan to Share IPD: No